CLINICAL TRIAL: NCT01008982
Title: A Phase 2, Proof of Concept, 52-Week Open Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B™), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects With Primary Sjögren's Syndrome.
Brief Title: Efficacy and Safety of Belimumab in Primary Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Udine (Other)
Collaborators: Azienda Ospedaliera S. Maria della Misericordia (Other)
Responsible Party: Principal Investigator, Salvatore De Vita, prof, MD, University of Udine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS-BEL-01-1.0
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Sjögren's Syndrome
Keywords: Belimumab,Sjögren's Syndrome.; Have a diagnosis of primary SS according to the updated American European Consensus Group Criteria
MeSH Terms: conditions — Sjogren's Syndrome | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental)
  Interventions: Drug: LimphoStat-B

INTERVENTIONS:
Drug: LimphoStat-B — subjects will receive 10 mg/kg belimumab, in solution for infusion, monthly
  Other Names: Belimumab

SUMMARY:
Background and rationale Sjögren's syndrome (SS) is a systemic autoimmune disease characterized by chronic inflammation of salivary and lachrymal glands, frequently accompanied by systemic symptoms. The presence of various autoantibodies such as rheumatoid factor (RF) and anti-SSA/SSB antibodies, as well as hypergammaglobulinemia, reflect B cell hyperactivity. About five percent of patients with SS develop malignant B cell lymphoma, usually of the mucosa-associated lymphoid tissue (MALT) type and most frequently located in the major salivary glands. Currently, there is a lack of evidence-based intervention therapy which may influence SS-related chronic inflammation and lymphoproliferation. B cells are involved in the pathogenesis of SS, and B cell downregulation may lead to a decrease of disease activity. Patients with more residual exocrine gland function, e.g., those with SS of shorter duration, might better benefit from systemic therapy, as reported in a preliminary study on the efficacy of B-cell depletion in SS.This study will examine the effect of the drug Belimumab in patients with SS. Patients aged more than 18 years with SS may be eligible for this study. Candidates will be screened with complete history and physical examination, chest x-rays, and oral and eye examinations.

DETAILED DESCRIPTION:
A Phase 2, proof of concept, 52 Week Open Study to Evaluate the Efficacy and Safety of Belimumab (HGS1006, LymphoStat-B), a Fully Human Monoclonal Anti-BLyS Antibody, in Subjects with Sjögren's Syndrome (pSS)

Clinical Development Phase: 2

A total of 15 patients will be recruited

Objectives

To evaluate the proof of concept of efficacy of belimumab in subjects with SS To evaluate the safety and tolerability of belimumab in subjects with SS

This is a Phase 2, proof of concept, 52-week open study to evaluate the efficacy and safety of belimumab in subjects with active SS. In addition to receiving standard stable therapy, subjects will receive 10 mg/kg belimumab. At week 28, if worsening any patient will exit the study band considered as a treatment failure.

If the disease is stable at week 28, and if both the referent clinician and the patient agree in continuing the study, the study will continue up to week 52 in that patient, since a delayed response may occur (as shown in systemic lupus erythematosus patients treated with belimumab: Chathman et al. Arthritis Rheumatism 2008 ).

Inclusion criteria

Have a diagnosis of primary SS according to the updated American European Consensus Group Criteria. In addition, patients must be always positive for anti-SSA or anti-SSB antibodies

Have the presence, at screening, of Systemic involvement (polysynovitis, skin, renal, lung, CNS involvement, peripheral neuropathy, vasculitis, autoimmune cytopenia, defined in Annex 1) or persistent (up to 2 months) parotid, submandibular or lachrymal gland swelling of more than 2 cm

OR

Objective sicca (positive oral and/or ocular tests reported in the American European Consensus Group Criteria) with at least one among the following biological features of serum B lymphocyte activation :

increased IgG levels increased free light chain levels of immunoglobulins (according to central laboratory ranges) increased serum beta2-microglobulin levels decreased C4 levels (C4 levels inferior to central laboratory ranges) monoclonal gammapathy cryoglobulinemia

OR

c) SS of more recent onset, i.e., less than 5 years of duration of symptoms, associated with: i) oral or ocular dryness and ii) fatigue and iii) musculoskeletal pain (i.e, 3 criteria for response as reported at page (ix-x), characterized by VAS score more than 50/100 in all the 3 fields.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age.
2. Have a diagnosis of primary SS according to the updated American European Consensus Group Criteria -

Exclusion Criteria:

1. Have received treatment with any BLyS-targeted (BLyS-receptor fusion protein [BR3], TACI Fc, or belimumab) at any time.
2. Have a Grade 3 or greater laboratory abnormality based on the protocol toxicity scale except for the following that are allowed:

   * Stable Grade 3 prothrombin time (PT) secondary to warfarin treatment.
   * Stable Grade 3/4 proteinuria (≤ 6 g/24 hour equivalent by spot urine protein to creatinine ratio allowed).
   * Stable Grade 3 neutropenia or stable Grade 3 white blood cell count

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the proof of concept of efficacy of belimumab in subjects with SS. To evaluate the safety and tolerability of belimumab in subjects with SS | week 28 and week 52

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore De Vita, MD, Principal Investigator — Rheumatology Clinic
Locations (1):
- Salvatore De Vita, Udine, Italy, Italy

REFERENCES:
- [Derived] Pontarini E, Fabris M, Quartuccio L, Cappeletti M, Calcaterra F, Roberto A, Curcio F, Mavilio D, Della Bella S, De Vita S. Treatment with belimumab restores B cell subsets and their expression of B cell activating factor receptor in patients with primary Sjogren's syndrome. Rheumatology (Oxford). 2015 Aug;54(8):1429-34. doi: 10.1093/rheumatology/kev005. Epub 2015 Mar 3. PMID 25740829